CLINICAL TRIAL: NCT01238562
Title: A Randomized, Open-label, Single-dose, Dose-escalation, Self-controlled Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of YPEG-Filgrastim in Cancer Patients Receiving Chemotherapy
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of YPEG-Filgrastim in Chemotherapy Patients
Acronym: Filgrastim
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: TB1004CSF
Record Dates: First submitted 2010-11-05; First posted 2010-11-10 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2010-03

CONDITIONS: Chemotherapy Patients
Keywords: cancer patient; chemotherapy; carboplatin; taxol; cyclophosphamide; pharmorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- YPEG-Filgrastim, 10mcg/kg (Experimental)
  Interventions: Drug: YPEG-Filgrastim
- YPEG-Filgrastim, 20mcg/kg (Experimental)
  Interventions: Drug: YPEG-Filgrastim
- YPEG-Filgrastim, 30mcg/kg (Experimental)
  Interventions: Drug: YPEG-Filgrastim
- YPEG-Filgrastim, 45mcg/kg (Experimental)
  Interventions: Drug: YPEG-Filgrastim
- YPEG-Filgrastim, 60mcg/kg (Experimental)
  Interventions: Drug: YPEG-Filgrastim

INTERVENTIONS:
Drug: YPEG-Filgrastim — s.c, single dose of 10mcg/kg of YPEG-Filgrastim at 48hr of cycle 2, followed by daily s.c either 2.5 mcg/kg or 5 mcg/kg of filgrastim(TOPNEUTER) starting from 48hr of cycle 3 until WBC≥10,000 per cubic milliliter or ANC≥5,000 per cubic milliliter in two continuous daily tests after ANC nadir.
  Arms: YPEG-Filgrastim, 10mcg/kg
Drug: YPEG-Filgrastim — s.c, single dose of 20mcg/kg of YPEG-Filgrastim at 48hr of cycle 2, followed by daily s.c either 2.5 mcg/kg or 5 mcg/kg of filgrastim(TOPNEUTER) starting from 48hr of cycle 3 until WBC≥10,000 per cubic milliliter or ANC≥5,000 per cubic milliliter in two continuous daily tests after ANC nadir.
  Arms: YPEG-Filgrastim, 20mcg/kg
Drug: YPEG-Filgrastim — s.c, single dose of 30mcg/kg of YPEG-Filgrastim at 48hr of cycle 2, followed by daily s.c either 2.5 mcg/kg or 5 mcg/kg of filgrastim(TOPNEUTER) starting from 48hr of cycle 3 until WBC≥10,000 per cubic milliliter or ANC≥5,000 per cubic milliliter in two continuous daily tests after ANC nadir.
  Arms: YPEG-Filgrastim, 30mcg/kg
Drug: YPEG-Filgrastim — s.c, single dose of 45mcg/kg of YPEG-Filgrastim at 48hr of cycle 2, followed by daily s.c either 2.5 mcg/kg or 5 mcg/kg of filgrastim(TOPNEUTER) starting from 48hr of cycle 3 until WBC≥10,000 per cubic milliliter or ANC≥5,000 per cubic milliliter in two continuous daily tests after ANC nadir
  Arms: YPEG-Filgrastim, 45mcg/kg
Drug: YPEG-Filgrastim — s.c, single dose of 60mcg/kg of YPEG-Filgrastim at 48hr of cycle 2, followed by daily s.c either 2.5 mcg/kg or 5 mcg/kg of filgrastim(TOPNEUTER) starting from 48hr of cycle 3 until WBC≥10,000 per cubic milliliter or ANC≥5,000 per cubic milliliter in two continuous daily tests after ANC nadir.
  Arms: YPEG-Filgrastim, 60mcg/kg

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics, pharmacodynamics of a single-dose of YPEG-Filgrastim in cancer patients receiving chemotherapy, and will establish dose-response relationships between YPEG-Filgrastim and Filgrastim(rhG-CSF, TOPNEUTER).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18～70yrs
* Signed informed consent
* Confirmed malignant tumor patients by histopathological or cytological diagnosis, suitable for chemotherapy with carboplatin combined with taxol or cyclophosphamide combined with pharmorubicin
* Karnofsky score ≥70
* Life expectancy >3 months
* WBC≥3,500 per cubic milliliter, ANC≥1,500 per cubic milliliter, PLT≥100,000 per cubic milliliter
* Normal coagulation function, no evidences of hemorrhage
* Normal liver, heart, kidney function

Exclusion Criteria:

* Pregnant or lactating females
* Proven active infectious diseases (e.g. viral hepatitis, TB)
* Not adequately controlled infections
* Known hypersensitivity to filgrastim or any other components of the study drug
* Unstable or uncontrolled cardiac disease or hypertension
* Currently participated in any other clinical trials
* Patients with previous or expected to receive systemic radiotherapy
* Evidence of metastatic disease in bone marrow, brain, et al
* Alcoholic or drug abusers
* Other conditions which in the opinion of the investigator preclude enrollment into the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Measurement of absolute neutrophil counts in the 3 cycles for pharmacodynamic study. | each cycle

SECONDARY OUTCOMES:
Measurement of serum concentration of drugs for Pharmacokinetic study. | each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuankai, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China